CLINICAL TRIAL: NCT03456986
Title: Improvements in Cognitive Skills of Older Adults Using Dynamic Visual Attention Training
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was never funded by NIH as anticipated.
Sponsor: Perception Dynamics Institute (Industry)
Collaborators: University of California, San Diego (Other); University of South Alabama (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1R43 AG059547-01
Record Dates: First submitted 2018-02-22; First posted 2018-03-07 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2018-04

CONDITIONS: Age Related Cognitive Decline

STUDY DESIGN:
Intervention Model Description: The feasibility of PATH neurotraining will be evaluated by comparing it with another cognitive training program, Brain HQ's Target Tracker, and ascertaining the relative advantage(s) of PATH neurotraining for enhancing cognition in older adults between 55 and 75 years of age whose cognition is either in the age-normative range or in the mild cognitive impairment (MCI) range of standardized psychometric measures.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: All data will be encrypted so participant's ID does not identify person. Two interventions, both improving motion discrimination will be investigated. Both have the potential of improving cognitive skills, so staff will not think one works better than the other. All data will be input by the senior research assistants who will not know what group a participant belonged to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PATH neurotraining (treatment) (Experimental): Subject looks at computer screen to determine whether bars in fish-shaped window move left or right relative to background bars. The subject reports which way center pattern moves by pushing left or right arrow key, receiving brief tone if incorrect. Program adaptively changes contrast of test pattern in order to keep subject at 79% correct. There are levels of difficulty introduced by making the background pattern more similar to that in fish, by increasing pattern's complexity level, and by increasing number of directions of movement from one to two directions of motion. Intervention will be trained for one training cycle, between 10-20 minutes, 3 times each week for 12 weeks.
  Interventions: Behavioral: PATH neurotraining
- Orientation Discrimination (control) (Active Comparator): Subject looks at computer screen to determine whether bars in center circular window are tilted left or right relative to vertically oriented background bars. The subject reports which way center pattern is tilted by pushing left or right arrow key, receiving brief tone if incorrect. Program adaptively changes orientation of test pattern in order to keep subject at 79% correct. There are levels of difficulty introduced by making the background pattern colored or black and white, and by increasing pattern's complexity level. This Intervention will be trained for one training cycle, between 10-20 minutes, 3 times each week for 12 weeks.
  Interventions: Behavioral: Orientation Discrimination

INTERVENTIONS:
Behavioral: PATH neurotraining — Tunes up the center of the motion discrimination (dorsal stream) working range
  Arms: PATH neurotraining (treatment)
Behavioral: Orientation Discrimination — Tunes up the ventral stream most sensitive to high contrast and colored patterns.
  Arms: Orientation Discrimination (control)

SUMMARY:
The proposed SBIR Phase I study tests the feasibility of PATH neurotraining for improving cognitive skills in older adults and, potentially, forestalling or protecting against cognitive decline and dementia. The feasibility of PATH neurotraining will be evaluated by comparing it with another cognitive training program, Brain HQ's Target Tracker, and ascertaining the relative advantage(s) of PATH neurotraining for enhancing cognition in older adults between 55 and 75 years of age whose cognition is either in the age-normative range or in the mild cognitive impairment (MCI) range of standardized psychometric measures. MEG/MRI source imaging will be used on 12 of the PATH group participants to determine whether the behavioral results are verified by improvements in the dorsal, attention, and executive control networks.

DETAILED DESCRIPTION:
The goal of this study is to show that neurotraining in the center of the motion working range (PATH) that improves the contrast sensitivity for direction discrimination (dorsal stream activity significantly improves cognitive skills in older adults more than in those who do training to improve orientation discrimination: ventral stream activity (sham training). Brain training will be administered for 20 minutes three times a week for 12 weeks: Arm 1) PATH neurotraining and Arm 2) Sham training. The investigators predict that older adults who do PATH neurotraining will improve their visual and cognitive skills, improving attention, multitasking, processing speed, reading fluency, and working memory, significantly more than those doing sham training. This prediction will be evaluated by measuring whether older adults improve on standardized tests of cognitive skills following PATH neurotraining more than older adults doing orientation discrimination training to improve processing speed and attention. MEG brain imaging will be used to show that PATH training improves the dorsal, attention, and executive control networks, as found previously, more than does sham training. The investigators predict these improvements will be found in both healthy adults and those with MCI.

The feasibility of rapid, effective brain training will be evaluated by using behavioral methods to remediate age-related cognitive decline, and to treat the cognitive impairment and/or behavioral symptoms associated with MCI, as well as to slow and/or reverse the course of cognitive decline or to prevent it entirely. PATH neurotraining provides a computer-based product to remediate the visual and cognitive difficulties of older adults rapidly and effectively. The innovative PATH neurotraining improves the center of the motion working range, whereas the sham training improves the center of the orientation discrimination working range. The two brain training groups will be balanced, in terms of healthy older adults and those with MCI. A subject will be considered to have MCI if the WAIS Working Memory Index score is less than 50 percent, and the MOCA has a score of 19-25. These groups will also be balanced in terms of age and reading speed, a sensitive measure of processing speed.

Half of the older adults will complete the PATH neurotraining for 12 weeks and half will complete sham training for 12 weeks. An additional 12 weeks will be needed to train staff, recruit subjects, and complete the standardized tests and MEG imaging. The choice of which adults will do each type of brain training will be randomized, to be determined by study statistician Prof. John Shelley-Tremblay. After initial standardized testing, 12 adults doing PATH training will be selected for pre-post MEG brain imaging.

Precise measurements using pre- and post- standardized tests of cognitive skills will be used to validate the improved visual and cognitive (attention, processing speed, and memory) performance reported previously in older adults. Standardized tests and MEG imaging on a subset will be administered by staff before and after cognitive training to evaluate improvements in cognitive skills following treatment (PATH neurotraining) and control (sham training) interventions.

Evaluating improvements in cognitive skills of older adults will be grouped by subject type: whether the adult is healthy or has MCI to determine which intervention improves cognitive skills the most. The investigators predict that PATH neurotraining will significantly improve (at p ≤ 0.05) reading speed, working memory and attention (cognitive flexibility) in older adults more than after training on sham training. This will be evaluated by both: 1) measuring whether older adults improve on the standardized tests listed above following brain training, and 2) MEG brain source imaging to validate that dorsal stream, attention, and executive control networks improve in function significantly following PATH neurotraining.

This study plans to study 40 older adults between the ages of 55 to 75, 20 in each group. Older adults will be recruited by posting brochures, getting referrals from Dr. James Brewer and Dr. Michael Lobatz, both who work with older adults having Alzheimer's Disease.

Training Procedures. Brain training exercises will be implemented in a high fidelity manner, using a detailed written protocol that all Research Assistants (RAs) are trained to follow meticulously, new PATH training movies and new motivational strategies. Staff will be hired at UCSD following interviews with Cognitive Science undergraduates who answered an advertisement on Handshake, the UCSD portal advertising for internships for UCSD students. Hiring RAs for this project and a Senior RA (SRA) to monitor study will be done by the PI at UCSD. Eleven RAs will be hired to administer standardized tests and both types of brain training to older adults at Perception Dynamics Institute (PDI) having a clinic ideal for collecting data in quiet surroundings with easy access for older adults. New training videos aimed at older adults will be developed by Leslie Peters at Desert Bay Productions in Encinitas.

The RAs will ensure each older adult is on task, completing the PATH neurotraining (pathtoreading.com) designed to activate the dorsal brain pathways and Sham training designed to activate the ventral brain pathways, and is progressing through each program in a timely manner by examining their data. The PI, having extensive experience conducting controlled validation studies, will be in charge of training all staff, running daily operations which requires supervising standardized testing and administering the interventions.

Measures To Evaluate Effectiveness of Training to Improve Visual and Cognitive Skills.

Behavioral Measure: Standardized testing of cognitive skills will be conducted at PDI by UCSD undergraduate Cognitive Science students trained by the PI, as done previously. All participants will undergo a review of their medical history and everyday activities impacted as they aged using a 9-item questionnaire described in Human Subjects. Since these are timed tests with test items not able to be memorized for future testing, practice effects are minimized. Cognitive assessments, which take about one hour to administer, will be evaluated before and after training by standardized tests for adults to measure:

1. Attention using Delis-Kaplan Executive Function System (D-KEFS) Color-Word Interference test (10 minutes).
2. Reading Speed using Computer-Based Reading Rate task (reading 6 words of text on screen) from interesting story at increasing speeds to measure 2 reading rate thresholds using a double-staircase procedure, after being trained by watching ReadingRate movie. (5 minutes).
3. Processing Speed Index (Wechsler Adult Intelligence Scale (WAIS)-4 Coding and Symbol Search subtests) and Working Memory Index (WAIS-4 Digit Span and Letter-Number Sequencing subtests), (10 minutes).
4. Visual Working Memory (VWM) using Test of Information Processing Skills, having two distractor tasks, a counting task and repeating a short sentence, having to animal names at end of test (10 minutes).

Biomarker Measure: MEG Imaging will be used to provide a Biomarker to show that only improving dorsal stream function improves cognitive skills in older adults. To establish the feasibility of PATH neurotraining to improve cognitive function in older adults, Prof. Ming-Xiong Huang will record voxel-wise MEG source magnitude images, from 12 older adults to determine the cortical areas improving in function following PATH neurotraining and following sham training. MEG brain imaging, using the Fast-VESTAL procedure (Huang et al. 2016, 2017, 2018), showed that this movement-discrimination training improved time-locked activity in the dorsal stream, attention, and executive control networks. MEG images covering the whole brain, for each frequency band, following the Fast-VESTAL procedure, to measure time-locked signals during a working memory N-back task will be used to evaluate improvements in brain function. The N-back task is one of the most frequently used WM paradigms (Gevins and Cutillo, 1993) to investigate the neural basis of WM processes. Two MEG exams will be performed for each participant, one before and another after the PATH or sham training.

N-back Working Memory Task. Participants will undergo MEG recordings while performing an N-back WM task. The task entails on-line monitoring, updating, and manipulation of remembered information. During the task, the participant is required to monitor a series of letters (both upper and lower case) presented for 500 ms in the middle of the screen. A fixation cross is presented during the 3000 ms interstimulus interval. The participant is instructed to respond only when a letter is presented that matches (i.e. target) the one presented n trials previously, while not to responding to the unmatched stimuli (non-target). Two load conditions will be used (1-back and 2-back), which place increasing demands on WM processes. About 50 trials per load condition will be collected for each participant. Performance will be recorded using an MEG-compatible response pad, in which index finger blocks-and-unblocks a laser-beam. The outputs of the response pad including reaction times will be recorded in the MEG file. The percent correct responses to target and non-target stimuli will be measured.

Different from the conventional MEG approach in which sensor waveforms are averaged with respect to the onset of the stimuli, the sensor covariance matrices for individual trials will be calculated. Then a total sensor-waveform covariance matrix of the target condition will be calculated by averaging across the covariance matrices from individual trials for the target stimuli. Then the covariance matrices across trials will be averaged. Using the total covariance matrix, voxel-wise MEG source magnitude images that cover the whole brain will be obtained for each subject, and each frequency band, following the Fast-VESTAL procedure, see Method in (Huang et al., 2014) and Appendix in (Huang et al., 2016), measuring time-locked signals during a working memory N-back task to evaluate improvements in brain function. An Objective Pre-whitening Method will be applied to remove correlated environmental noise and objectively select the dominant eigen-modes of sensor-waveform covariance matrix (Huang et al., 2014).

Another goal is to study the neuronal correlates of potential cognitive dysfunctions observed using behavioral measures in older adults. Voxel-wise correlation analyses will also be performed to examine the association of N-back source images and neuropsychological scores. All subjects will be combined together for the correlation analyses. In each frequency band, the MEG source images in the MNI-152 space (following the spatial smoothing and logarithm transformation) will be formed into three 4D data sets: Dimensions 1-3 represent the x-, y-, and z-coordinates, and the fourth dimension represents all subjects. A total of eight data sets will be created for 1- and 2-back conditions, and for four frequency bands. Next, along the fourth dimension, voxel-wise repeated measure correlation analyses (Bakdash and Marusich, 2017) will be performed between MEG source images and each of the neuropsychological scores. For each frequency band, the 1- and 2-back conditions will be treated as repeated measures in such analyses. In this study, we will only examine the neuropsychological scores that show statistical group differences. The repeated measure correlation analyses creates r-value correlation maps, and cluster analysis that will be used to control for family-wise errors at a corrected p<0.01 level for the r-value maps, similar to the correction procedure for the F-value maps.

ELIGIBILITY:
Inclusion Criteria:

* All older adults who want to participate and can do the intervention tasks, agree to the time commitment, and are not excluded for reasons cited below

Exclusion Criteria:

* Have severe depressions or suicidal thoughts or tendencies
* Have had a stroke, Traumatic Brain Injury, or metabolic derangements causing cognitive impairments, such as alcohol or substance abuse.
* Cannot complete the PATH neurotraining task, pushing the left or right arrow key on the computer after moving patterns are presented briefly on the computer screen will be excluded. That has never been a problem previously, so we do not anticipate excluding anyone for this reason.
* Cannot drive to the test site, eliminating those with major functional issues in cognition.
* Have been given a diagnosis of dementia by their doctor.
* Do not agree to complete the study after hearing the time commitment involved.
* For the MEG portion of study, have extensive metal dental hardware )e.g. braces and large metal dentures; fillings are acceptable) or other metal objects in the head, neck, or face areas that cause artifacts in the MEG data, not removable during pre-processing

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09-04 (Estimated); Primary Completion 2019-04-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Reading Speed | 12 weeks (before and after intervention training)
  Number of words/minute subject can read 6 words of text from interesting story. Measures improvements in processing speed.

SECONDARY OUTCOMES:
Auditory Working Memory | 12 weeks (before and after intervention training)
  The WAIS Working Memory Index Standardized Percentile Rank that goes from < 0.1% to > 99.9%
Visual Working Memory | 12 weeks (before and after intervention training)
  The Test of Information Processing Skills Visual Working Memory Standardized Percentile Rank that goes from < 1% to > 99%
Attention | 12 weeks (before and after intervention training)
  DKEFS Color-Word Interference Test standardized scores for Inhibition Scaled Scores that go from 1 to 19 converted to Standardized Percentile Rank from 0.5% to 99.9%
Attention Switching | 12 weeks (before and after intervention training)
  DKEFS Color-Word Interference Test standardized scores for Inhibition Switching Scaled Scores that go from 1 to 19 converted to Standardized Percentile Rank from 0.5% to 99.9%
Processing Speed | 12 weeks (before and after intervention training)
  WAIS Processing Speed Index Standardized Percentile Rank that goes from < 0.1% to > 99.9%
DLPFC Function | 12 weeks (before and after intervention training)
  Using the total covariance matrix, voxel-wise MEG source magnitude images that cover the whole brain will be obtained for each subject, and each frequency band, following the Fast-VESTAL procedure, measuring time-locked signals during a working memory N-back task to evaluate improvements in brain function in DLPFC (working memory).
ACC Function | 12 weeks (before and after intervention training)
  Using the total covariance matrix, voxel-wise MEG source magnitude images that cover the whole brain will be obtained for each subject, and each frequency band, following the Fast-VESTAL procedure, measuring time-locked signals during a working memory N-back task to evaluate improvements in brain function in ACC (attention network).
Precuneus/PCC | 12 weeks (before and after intervention training)
  Using the total covariance matrix, voxel-wise MEG source magnitude images that cover the whole brain will be obtained for each subject, and each frequency band, following the Fast-VESTAL procedure, measuring time-locked signals during a working memory N-back task to evaluate improvements in brain function in Precuneus/PCC (attention network).

CONTACTS AND LOCATIONS:
Overall Officials: Teri Lawton, PhD, Principal Investigator — Perception Dynamics Institute
Locations (2):
- United States (2):
  - UCSD Radiology Laboratory, La Jolla, California
  - Perception Dynamics Institute, Solana Beach, California

IPD SHARING:
Plan to Share IPD: Yes
After completion of the study, deidentified data will be made available to qualified outside investigators following NIH Data Sharing guidelines; none of the data will be considered proprietary. Most of the data for this study will be collected through standardized tests of attention, processing speed, and working memory to be administered by the staff on this project.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: May 2019 for 10 years.
Access Criteria: Qualified investigator